CLINICAL TRIAL: NCT02475655
Title: A Randomized, Pilot Study of Ruxolitinib in Antiretroviral-Treated HIV-Infected Adults
Brief Title: Evaluating the Safety and Tolerability of Ruxolitinib in Antiretroviral-Treated HIV-Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5336; 11977 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2015-06-16; First posted 2015-06-19 (Estimated); Results first posted 2019-04-18 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Ruxolitinib (Experimental): Participants received ruxolitinib twice a day for 5 weeks. Participants were required to remain on ART regimen (not provided by the study) for the duration of the study.
  Interventions: Drug: Ruxolitinib
- Arm B: No Study Treatment (No Intervention): Participants did not receive any study treatment. Participants were required to remain on ART regimen (not provided by the study) for the duration of the study.

INTERVENTIONS:
Drug: Ruxolitinib — 10 mg orally twice daily for 5 weeks
  Arms: Arm A: Ruxolitinib

SUMMARY:
The purpose of this study was to evaluate the safety and tolerability of ruxolitinib in HIV-positive adults who were virologically suppressed and who were on antiretroviral therapy (ART).

DETAILED DESCRIPTION:
Ruxolitinib is a medication approved by the U.S. Food and Drug Administration (FDA) to treat myelofibrosis, a disorder in which bone marrow is replaced by scar (fibrosis) tissue. Many of the cytokines affected by myelofibrosis are also affected by HIV. Because of this, ruxolitinib may also be a possible treatment for HIV. The purpose of this study was to evaluate the safety and tolerability of ruxolitinib in HIV-positive adults who were on ART and who were virologically suppressed. Researchers evaluated the effect ruxolitinib had on inflammation and immune activation.

This study enrolled HIV-positive adults who were on select ART regimens and who had viral suppression. ART was not provided by the study; participants continued to receive ART from their own health care providers. Participants were randomly assigned to receive either ruxolitinib (Arm A) or no study treatment (Arm B) in 2:1 ratio. Participants in Arm A received ruxolitinib twice a day for 5 weeks. All participants attended study visits at entry (Day 0) and Weeks 1, 2, 4, 5, 10, and 12. These visits included physical examinations, clinical assessments, blood collection, adherence assessments, oral swab collection, and pregnancy testing for female participants. At Weeks 1 and 4, participants in Arm A took part in pharmacokinetic (PK) sampling, which involved having blood drawn several times over 6 to 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* CD4+ T cell count greater than 350 cells/mm^3 within 45 days prior to study entry
* Documented virologic suppression defined as HIV-1 RNA level below the limit of quantification (eg, less than 40, less than 50, or less than 75 copies/mL, depending on the assay) using an FDA-approved assay with a quantification limit of 75 copies/mL or lower for at least 48 weeks prior to study entry
* Screening HIV-1 RNA level below the limit of quantification
* Tuberculosis (TB) screening within 365 days of the screening visit diagnosed by tuberculin skin test or interferon gamma release assay
* Currently on continuous ART for at least 730 days prior to study entry, defined as continuous ART for the 730 days period, inclusive, prior to study entry with no ART interruption longer than 7 consecutive days. NOTE: The current regimen must include TDF/FTC, TAF/FTC, TDF+3TC, or ABC/3TC; plus a nonnucleoside reverse transcriptase inhibitor or integrase strand transfer inhibitor (NNRTI or INSTI, not containing cobicistat) for at least 60 days, inclusive, prior to study entry.
* The following laboratory values obtained within 45 days prior to entry:

  * Absolute neutrophil count (ANC) greater than or equal to 1,000/mm^3
  * Hemoglobin greater than 12.0 g/dL for men and greater than 11.0 g/dL for women
  * Platelets greater than or equal to 140,000/mm^3
  * Calculated creatinine clearance (CrCl) greater than or equal to 70 mL/min (by Cockcroft Gault equation)
  * Aspartate aminotransferase (AST) (SGOT) less than or equal to 1.5x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) (SGPT) less than or equal to 1.5x ULN
  * Alkaline phosphatase less than or equal to 1.5x ULN
* For females of reproductive potential, a negative serum or urine pregnancy test with a sensitivity of 25 mIU/mL within 72 hours, inclusive, prior to study entry
* All participants must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization)
* All participants of reproductive potential, who were participating in sexual activity that could lead to pregnancy, must agree to use at least one reliable method of contraception while receiving the study drugs and for 7 weeks after stopping the medications
* Ability and willingness of participant or legal representative to provide written informed consent and attend study visits as scheduled at a participating site

Exclusion Criteria:

* A current or past history of progressive multifocal leukoencephalopathy
* Breastfeeding or pregnancy
* Use of strong inhibitors or inducers of CYP3A4 including a protease inhibitor, cobicistat or entry inhibitors as part of the current ART regimen or other concomitant therapy
* Known allergy/sensitivity or any hypersensitivity to components of study drug or their formulation
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Acute or serious illness or infection requiring systemic treatment and/or hospitalization within 60 days prior to entry
* Vaccinations (other than influenza) less than or equal to 45 days prior to the study entry visit.
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), systemic cytotoxic chemotherapy or investigational therapy less than or equal to 60 days prior to study entry
* Any current diagnosis or past history of a significant cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, neuropsychiatric, psychiatric, or other serious illness that, in the opinion of the investigator, could constitute a risk when taking investigational product or could interfere with the interpretation of data or affect the participant's ability to participate in the study. Diagnoses that would lead to exclusion include, but were not limited to the following:

  * CDC category C AIDS-indicator conditions
  * NOTE A: Except HIV encephalopathy, HIV wasting, esophageal candidiasis, or pneumocystis pneumonia without dissemination.
  * NOTE B: List available: http://www.cdc.gov/mmwr/preview/mmwrhtml/00018871.htm
  * Herpes zoster (dermatomal or non-dermatomal).
  * NOTE C: A history of prior chickenpox was not exclusionary.
  * Lymphoproliferative malignancy
  * Chronic liver disease of any etiology and any degree of severity
  * Chronic hepatitis, except for hepatitis C that has been cured (defined as a Sustained Virologic Response, which is an undetectable HCV-RNA at 12 weeks or more after completing treatment measured by a sensitive, qualitative, or quantitative HCV-RNA assay)
  * Disseminated fungal infection of any type or duration that is not limited to cutaneous or mucocutaneous surfaces
  * A medical disorder that predisposes to bleeding
* Change in the ART regimen within 12 weeks, inclusive, prior to study entry or intended modification of ART during the study.
* History of untreated latent tuberculosis infection (LTBI) diagnosed by tuberculin skin test or interferon gamma release assay. LTBI treatment would consist of 9 months of isoniazid or an equivalent therapy completed at least 4 weeks prior to study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2018-02-18 (Actual); Study Completion 2018-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Marconi, MD, Study Chair — Emory University; Jeffrey Lennox, MD, Study Chair — Emory University
Locations (14):
- United States (14):
  - Alabama CRS, Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - Northwestern University CRS, Chicago, Illinois
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - Weill Cornell Chelsea CRS, New York, New York
  - Weill Cornell Uptown CRS, New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS, Rochester, New York
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - Case Clinical Research Site, Cleveland, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - The Miriam Hospital Clinical Research Site (TMH CRS) CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee

REFERENCES:
- [Derived] Marconi VC, Moser C, Gavegnano C, Deeks SG, Lederman MM, Overton ET, Tsibris A, Hunt PW, Kantor A, Sekaly RP, Tressler R, Flexner C, Hurwitz SJ, Moisi D, Clagett B, Hardin WR, Del Rio C, Schinazi RF, Lennox JJ. Randomized Trial of Ruxolitinib in Antiretroviral-Treated Adults With Human Immunodeficiency Virus. Clin Infect Dis. 2022 Jan 7;74(1):95-104. doi: 10.1093/cid/ciab212. PMID 33693561
- See also: DAIDS AE Grading Table, Version 2.0, November 2014 — https://rsc.niaid.nih.gov/sites/default/files/daids-ae-grading-table-v2-nov2014.pdf
- See also: Version 2.0 of the DAIDS EAE Manual — https://rsc.niaid.nih.gov/sites/default/files/manual-exped-aes-v2_0.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in 05/2016 and completed in 01/2018. Of N=119 screened subjects, N=60 were enrolled from fourteen clinical research sites in the United States.
Pre-assignment Details: Enrollment was stratified based on whether a participant was on an EFV-containing regimen.
Period: Overall Study
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Started | 40 | 20
Completed | 40 | 19
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [45 to 54] | 43.5 [31 to 54] | 49 [36.5 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 32 | 16 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 2 participants were missing race/ethnicity.
  Participants
    Race/Ethnicity: number analyzed (Participants) | 38 | 20 | 58
    Race/Ethnicity: White Non-Hispanic | 14 | 7 | 21
    Race/Ethnicity: Black Non-Hispanic | 19 | 10 | 29
    Race/Ethnicity: Hispanic (Regardless of Race) | 4 | 2 | 6
    Race/Ethnicity: More than One Race | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 20 | 60
Weight [Median (Inter-Quartile Range); unit: kg] | 89.2 [77.7 to 110.1] | 91.0 [76.1 to 104.5] | 89.2 [76.7 to 108.8]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 29.2 [25.0 to 33.5] | 29.5 [26.8 to 35.4] | 29.2 [25.6 to 34.3]
Entry CD4 Count [Median (Inter-Quartile Range); unit: cells/mm^3] | 798 [628 to 973] | 737 [610 to 930] | 791 [622 to 972]
Baseline CD4 Count [Median (Inter-Quartile Range); unit: cells/mm^3] — Baseline is the average of a participants Pre-entry and Entry measures. The median of all participant averages is reported.
  cells/mm^3 | 816 [639 to 958] | 855 [629 to 948] | 844 [639 to 948]
HIV-1 RNA [Count of Participants; unit: Participants]
  <40 copies/mL | 39 | 20 | 59
  >=40 copies/mL | 1 | 0 | 1
Baseline Interleukin 6 (IL-6) [Mean (Standard Deviation); unit: pg/mL] — Baseline is the geometric mean of a participants Pre-entry and Entry measures. The mean of all participant geometric means is reported. Population: Only reported in the as-treated population (had data at baseline and week 4/5; for the Ruxolitinib arm, remained on study treatment through week 4/5 and missed no more than 6 doses cumulatively; did not change ART, use prohibited medications, or have confirmed virologic failure through week 4/5; not found to be ineligible after randomization).
  pg/mL
    number analyzed (Participants) | 37 | 18 | 55
    (all) | 1.90 (1.84) | 1.69 (1.68) | 1.83 (1.79)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants on the Ruxolitinib Arm Who Experienced Any Safety Milestone Events While On-Treatment
Description: Events defined as safety milestones are listed below and together makeup the composite endpoint.
  * Confirmed CD4+ decline > 33% of entry and to < 350 cell/mm^3 (for participants with entry CD4+ T cell count < 700 cells/mm^3)
  * Confirmed CD4+ decline > 50% of entry (for participants with entry CD4+ T cell count ≥ 700 cells/mm^3)
  * Confirmed HIV-1 RNA level above the lower limit of quantification in the absence of an interruption of ART
  * New or recurrent CDC category C AIDS-indicator condition
  * HIV-1 associated infection including Herpes zoster
  * Lymphoproliferative malignancies
  * Grade 4 or recurrence of Grade 3 anemia/neutropenia
  * New diagnosis of pneumonia, sepsis, or bacteremia
  * Discontinuation of Ruxolitinib due to thrombocytopenia
  * Any Grade 4 or recurrence of Grade 3 toxicity related to study drug
  Percent experiencing a safety milestone will be reported.
Time Frame: Entry to Week 5
Population: Analysis was done on participants on the Ruxolitinib arm in the safety analysis population. These were all participants randomized to the Ruxolitinib arm who took at least one dose of Ruxolitinib.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Ruxolitinib
Number analyzed (Participants) | 40
percentage of participants | 2.5

2. Primary Outcome: Percentage of Participants Who Experienced Any Safety Milestones On-study From Entry to Week 5
Description: Events defined as safety milestones are listed below and together makeup the composite endpoint.
  * Confirmed CD4+ decline > 33% of entry and to < 350 cell/mm^3 (for participants with entry CD4+ T cell count < 700 cells/mm^3)
  * Confirmed CD4+ decline > 50% of entry (for participants with entry CD4+ T cell count ≥ 700 cells/mm^3)
  * Confirmed HIV-1 RNA level above the lower limit of quantification in the absence of an interruption of ART
  * New or recurrent CDC category C AIDS-indicator condition
  * HIV-1 associated infection including Herpes zoster
  * Lymphoproliferative malignancies
  * Grade 4 or recurrence of Grade 3 anemia/neutropenia
  * New diagnosis of pneumonia, sepsis, or bacteremia
  * Occurrence of Grade 2 or higher thrombocytopenia
  * Any Grade 4 or recurrence of Grade 3 toxicity
  Percent experiencing a safety milestone will be reported.
Time Frame: Entry to Week 5
Population: Analysis was done in the safety analysis population. The safety analysis population includes all participants randomized to the No Study Treatment arm and all participants who took at least one dose of Ruxolitinib among those randomized to the Ruxolitinib arm.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
percentage of participants | 2.5 | 0
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the percentage of participants experiencing safety milestones from Entry to Week 5; Test type: Superiority; p = 0.67, Fisher Exact — Not adjusted for multiple comparisons. One-sided 5% alpha; Fisher's Exact Mid P-Value

3. Primary Outcome: Percentage of Participants Who Experienced Each Safety Milestone That Occurred On-study From Entry to Week 5
Description: Events defined as safety milestones are listed below.
  * Confirmed CD4+ decline > 33% of entry and to < 350 cell/mm^3 (for participants with entry CD4+ T cell count < 700 cells/mm^3)
  * Confirmed CD4+ decline > 50% of entry (for participants with entry CD4+ T cell count ≥ 700 cells/mm^3)
  * Confirmed HIV-1 RNA level above the lower limit of quantification in the absence of an interruption of ART
  * New or recurrent CDC category C AIDS-indicator condition
  * HIV-1 associated infection including Herpes zoster
  * Lymphoproliferative malignancies
  * Grade 4 or recurrence of Grade 3 anemia/neutropenia
  * New diagnosis of pneumonia, sepsis, or bacteremia
  * Occurrence of Grade 2 or higher thrombocytopenia
  * Any Grade 4 or recurrence of Grade 3 toxicity
  Percent experiencing each safety milestone will be reported. Safety milestone categories are not mutually exclusive.
Time Frame: Entry to Week 5
Population: Analysis was done in the safety population. The safety analysis population includes all participants randomized to the No Study Treatment arm and all participants who took at least one dose of Ruxolitinib among those randomized to the Ruxolitinib arm.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
percentage of participants
  Confirmed CD4+ decline > 33% of entry | 0 | 0
  Confirmed CD4+ decline > 50% of entry | 0 | 0
  Confirmed HIV-1 RNA level above the lower limit | 0 | 0
  New/recurrent category C AIDS-indicator condition | 0 | 0
  HIV-1 associated infection including Herpes zoster | 0 | 0
  Lymphoproliferative malignancies | 0 | 0
  Grade 4/ recurrence of Grade 3 anemia/neutropenia | 0 | 0
  New diagnosis of pneumonia, sepsis, or bacteremia | 2.5 | 0
  Occurrence of Grade 2 or higher thrombocytopenia | 0 | 0
  Any Grade 4 or recurrence of Grade 3 toxicity | 0 | 0

4. Primary Outcome: Number of Participants With Premature Discontinuation of Study Treatment in the Ruxolitinib Arm
Description: Number of participants with premature discontinuation of study treatment are summarized.
Time Frame: Entry to Week 5
Population: All participants on the Ruxolitinib arm are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ruxolitinib
Number analyzed (Participants) | 40
Participants | 3

5. Primary Outcome: Fold Change in the Level of Plasma Interleukin 6 (IL-6) From Baseline to Week 4/5
Description: All values were log10 transformed prior to calculating change and conducting analyses and back transformed for presentation.
  Baseline is defined as the geometric mean of the Pre-entry and Entry values. Week 4/5 is defined as the geometric mean of the Week 4 and Week 5 values. Fold change was calculated as the value at Week 4/5 divided by the value at Baseline.
Time Frame: Pre-entry, Entry, Weeks 4 and 5
Population: Analysis was done in the as-treated population (had data at baseline and week 4/5; for the Ruxolitinib arm, remained on study treatment through week 4/5 and missed no more than 6 doses cumulatively; did not change ART, use prohibited medications, or have confirmed virologic failure through week 4/5; not found to be ineligible after randomization).
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 37 | 18
Fold Change | 0.93 [0.82 to 1.06] | 1.10 [0.84 to 1.44]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Plasma Interleukin 6 (IL-6) from baseline to week 4/5; Test type: Superiority; p = 0.18, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.85, 90% CI 2-sided [0.69 to 1.04] — Mean difference is Ruxolitinib geometric mean minus No Study Treatment geometric mean. All values were log10 transformed prior to calculating change and conducting analyses and back transformed for presentation

6. Secondary Outcome: Percentage of Participants on the Ruxolitinib Arm Who Experienced Any Safety Milestone Events During Total Follow-up
Description: as for outcome 1
Time Frame: Entry to Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Ruxolitinib
Number analyzed (Participants) | 40
percentage of participants | 7.5

7. Secondary Outcome: Percentage of Participants Who Experienced Any Safety Milestones On-study From Entry to Week 12
Description: as for outcome 2
Time Frame: Entry to Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
percentage of participants | 7.5 | 0
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the percentage of participants experiencing safety milestones from Entry to Week 12; Test type: Superiority; p = 0.40, Fisher Exact — Not adjusted for multiple comparisons. One-sided 5% alpha; Fisher's Exact Mid P-Value

8. Secondary Outcome: Percentage of Participants Who Experienced Each Safety Milestone That Occurred On-study From Entry to Week 12
Description: Events defined as safety milestones are listed below.
  * Confirmed CD4+ decline > 33% of entry and to < 350 cell/mm3 (for participants with entry CD4+ T cell count < 700 cells/mm3)
  * Confirmed CD4+ decline > 50% of entry (for participants with entry CD4+ T cell count ≥ 700 cells/mm3)
  * Confirmed HIV-1 RNA level above the lower limit of quantification in the absence of an interruption of ART
  * New or recurrent CDC category C AIDS-indicator condition
  * HIV-1 associated infection including Herpes zoster
  * Lymphoproliferative malignancies
  * Grade 4 or recurrence of Grade 3 anemia/neutropenia
  * New diagnosis of pneumonia, sepsis, or bacteremia
  * Occurrence of Grade 2 or higher thrombocytopenia
  * Any Grade 4 or recurrence of Grade 3 toxicity
  Percent experiencing each safety milestone will be reported. Safety milestone categories are not mutually exclusive.
Time Frame: Entry to Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
percentage of participants
  Confirmed CD4+ decline > 33% of entry | 0 | 0
  Confirmed CD4+ decline > 50% of entry | 2.5 | 0
  Confirmed HIV-1 RNA level above the lower limit | 2.5 | 0
  New/recurrent category C AIDS-indicator condition | 0 | 0
  HIV-1 associated infection including Herpes zoster | 0 | 0
  Lymphoproliferative malignancies | 0 | 0
  Grade 4/ recurrence of Grade 3 anemia/neutropenia | 0 | 0
  New diagnosis of pneumonia, sepsis, or bacteremia | 2.5 | 0
  Occurrence of Grade 2 or higher thrombocytopenia | 0 | 0
  Any Grade 4 or recurrence of Grade 3 toxicity | 0 | 0

9. Secondary Outcome: Number of Participants Who Experienced a Protocol-defined Reportable Adverse Event at Any Post-entry Time Point.
Description: Protocol-defined reportable adverse events include: all diagnoses regardless of grade, Grade 3 or higher sign/symptoms or laboratory values, any signs/symptoms or laboratory values that led to a change in treatment or met ICH, EAE, or SAE guidelines. See the Protocol Section References for links to the EAE manual.
  This is a subset of the events reported in the Adverse Events section.
Time Frame: Entry to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
Participants | 10 | 2

10. Secondary Outcome: Creatinine Clearance
Description: Creatinine clearance was calculated using the Cockcroft Gault equation. The arithmetic mean for each participant was calculated at week 1 and week 2 combined, week 4 and week 5 combined, and week 10 and week 12 combined.
Time Frame: Entry, Weeks 1, 2, 4, 5, 10, and 12
Population: Analysis was done in the safety analysis population for participants with available data. The safety analysis population includes all participants randomized to the No Study Treatment arm and all participants who took at least one dose of Ruxolitinib among those randomized to the Ruxolitinib arm.
Measure: Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
mL/min
  Entry | 118.5 [107.8 to 129.1] | 134.5 [115.4 to 153.6]
  Week 1/2: number analyzed (Participants) | 40 | 19
  Week 1/2 | 116.3 [106.6 to 126.0] | 130.2 [110.3 to 150.1]
  Week 4/5: number analyzed (Participants) | 40 | 19
  Week 4/5 | 117.3 [106.3 to 128.3] | 130.9 [111.5 to 150.4]
  Week 10/12: number analyzed (Participants) | 40 | 19
  Week 10/12 | 117.8 [108.3 to 127.2] | 126.6 [107.4 to 145.9]

11. Secondary Outcome: Change in Creatinine Clearance Values From Entry
Description: Creatinine clearance was calculated using the Cockcroft Gault equation. The arithmetic mean for each participant was calculated at week 1 and week 2 combined, week 4 and week 5 combined, and week 10 and week 12 combined.
  Absolute change was calculated as the value at Week 1/2 minus the value at Entry, the value at Week 4/5 minus the value at Entry, and the value at Week 10/12 minus the value at Entry.
Time Frame: Entry, Weeks 1, 2, 4, 5, 10, and 12
Population: Analysis was done in the safety analysis population for participants with results available at entry and at the follow-up time point. The safety analysis population includes all participants randomized to the No Study Treatment arm and all participants who took at least one dose of Ruxolitinib among those randomized to the Ruxolitinib arm.
Measure: Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
mL/min
  Change From Entry to Week 1/2: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 1/2 | -2.16 [-5.97 to 1.65] | -3.47 [-9.34 to 2.40]
  Change From Entry to Week 4/5: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 4/5 | -1.17 [-6.00 to 3.66] | -2.78 [-8.81 to 3.24]
  Change From Entry to Week 10/12: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 10/12 | -0.71 [-5.07 to 3.65] | -7.06 [-13.1 to -1.04]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in creatinine clearance from Entry to Week 1/2; Test type: Superiority; p = 0.70, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.31, 90% CI 2-sided [-4.27 to 6.90] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in creatinine clearance from Entry to Week 4/5; Test type: Superiority; p = 0.69, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.61, 90% CI 2-sided [-5.06 to 8.29] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 3: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in creatinine clearance from Entry to 10/12; Test type: Superiority; p = 0.09, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 6.35, 90% CI 2-sided [0.16 to 12.5]

12. Secondary Outcome: Creatinine
Description: The arithmetic mean for each participant was calculated at week 1 and week 2 combined, week 4 and week 5 combined, and week 10 and week 12 combined.
Time Frame: Entry, Weeks 1, 2, 4, 5, 10, and 12
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
mg/dL
  Entry | 0.99 [0.93 to 1.05] | 0.92 [0.85 to 0.99]
  Week 1/2: number analyzed (Participants) | 40 | 19
  Week 1/2 | 1.0 [0.94 to 1.06] | 0.95 [0.87 to 1.03]
  Week 4/5: number analyzed (Participants) | 40 | 19
  Week 4/5 | 1.01 [0.94 to 1.07] | 0.95 [0.87 to 1.02]
  Week 10/12: number analyzed (Participants) | 40 | 19
  Week 10/12 | 0.99 [0.93 to 1.04] | 0.99 [0.91 to 1.06]

13. Secondary Outcome: Change in Creatinine Values From Entry
Description: The arithmetic mean for each participant was calculated at week 1 and week 2 combined, week 4 and week 5 combined, and week 10 and week 12 combined.
  Absolute change was calculated as the value at Week 1/2 minus the value at Entry, the value at Week 4/5 minus the value at Entry, and the value at Week 10/12 minus the value at Entry.
Time Frame: Entry, Weeks 1, 2, 4, 5, 10, and 12
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
mL/min
  Change From Entry to Week 1/2: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 1/2 | 0.01 [-0.02 to 0.05] | 0.03 [-0.01 to 0.07]
  Change From Entry to Week 4/5: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 4/5 | 0.02 [-0.02 to 0.05] | 0.03 [-0.02 to 0.07]
  Change From Entry to Week 10/12: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 10/12 | -0.00 [-0.04 to 0.03] | 0.07 [0.03 to 0.10]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in creatinine from Entry to Week 1/2; Test type: Superiority; p = 0.58, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.02, 90% CI 2-sided [-0.06 to 0.03] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in creatinine from Entry to Week 4/5; Test type: Superiority; p = 0.79, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.01, 90% CI 2-sided [-0.06 to 0.04] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 3: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in creatinine from Entry to 10/12; Test type: Superiority; p = 0.016, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.07, 90% CI 2-sided [-0.11 to -0.02] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

14. Secondary Outcome: Absolute Neutrophil Count (ANC)
Description: as for outcome 12
Time Frame: Entry, Weeks 1, 2, 4, 5, 10, and 12
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
cells/mm^3
  Entry | 3558 [3049 to 4068] | 2730 [2244 to 3216]
  Week 1/2: number analyzed (Participants) | 40 | 19
  Week 1/2 | 3390 [2879 to 3901] | 3312 [2583 to 4041]
  Week 4/5: number analyzed (Participants) | 40 | 18
  Week 4/5 | 3307 [2834 to 3780] | 3163 [2434 to 3891]
  Week 10/12: number analyzed (Participants) | 40 | 19
  Week 10/12 | 3857 [3252 to 4462] | 3067 [2494 to 3639]

15. Secondary Outcome: Change in Absolute Neutrophil Count (ANC) Values From Entry
Description: as for outcome 13
Time Frame: Entry, Weeks 1, 2, 4, 5, 10, and 12
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
cells/mm^3
  Change From Entry to Week 1/2: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 1/2 | -169 [-476 to 138.9] | 510 [-11.6 to 1032]
  Change From Entry to Week 4/5: number analyzed (Participants) | 40 | 18
  Change From Entry to Week 4/5 | -251 [-506 to 3.70] | 400 [-233 to 1033]
  Change From Entry to Week 10/12: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 10/12 | 299 [-29.7 to 627] | 265 [-280 to 810]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in absolute neutrophil count (ANC) from Entry to Week 1/2; Test type: Superiority; p = 0.018, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -679, 90% CI 2-sided [-1146 to -212] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in absolute neutrophil count (ANC) from Entry to Week 4/5; Test type: Superiority; p = 0.021, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -651, 90% CI 2-sided [-1110 to -192] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 3: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in absolute neutrophil count (ANC) from Entry to Week 10/12; Test type: Superiority; p = 0.91, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 33.6, 90% CI 2-sided [-461 to 528] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

16. Secondary Outcome: Hemoglobin
Description: as for outcome 12
Time Frame: Entry, Weeks 1, 2, 4, 5, 10, and 12
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
g/dL
  Entry | 14.3 [13.8 to 14.8] | 14.3 [13.8 to 14.7]
  Week 1/2: number analyzed (Participants) | 40 | 19
  Week 1/2 | 14.0 [13.6 to 14.4] | 14.1 [13.6 to 14.7]
  Week 4/5: number analyzed (Participants) | 40 | 19
  Week 4/5 | 13.6 [13.2 to 14.1] | 14.2 [13.6 to 14.8]
  Week 10/12: number analyzed (Participants) | 40 | 19
  Week 10/12 | 14.4 [13.7 to 15.0] | 14.2 [13.7 to 14.7]

17. Secondary Outcome: Change in Hemoglobin Values From Entry
Description: as for outcome 13
Time Frame: Entry, Weeks 1, 2, 4, 5, 10, and 12
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
g/dL
  Change From Entry to Week 1/2: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 1/2 | -0.28 [-0.48 to -0.08] | -0.15 [-0.44 to 0.14]
  Change From Entry to Week 4/5: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 4/5 | -0.65 [-0.88 to -0.42] | -0.10 [-0.39 to 0.20]
  Change From Entry to Week 10/12: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 10/12 | -0.07 [-0.58 to 0.73] | -0.08 [-0.35 to 0.19]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in hemoglobin from Entry to Week 1/2; Test type: Superiority; p = 0.45, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.13, 90% CI 2-sided [-0.42 to 0.15] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in hemoglobin from Entry to Week 4/5; Test type: Superiority; p = 0.005, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.55, 90% CI 2-sided [-0.87 to -0.23] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 3: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in hemoglobin from Entry to Week 10/12; Test type: Superiority; p = 0.75, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.15, 90% CI 2-sided [-0.65 to 0.95] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

18. Secondary Outcome: Platelet Count
Description: as for outcome 12
Time Frame: Entry, Weeks 1, 2, 4, 5, 10, and 12
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: Platelets/mm^3
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
Platelets/mm^3
  Entry: number analyzed (Participants) | 40 | 19
  Entry | 238508 [222160 to 254855] | 261868 [237968 to 285769]
  Week 1/2: number analyzed (Participants) | 40 | 19
  Week 1/2 | 281525 [261316 to 301734] | 264492 [233571 to 295413]
  Week 4/5: number analyzed (Participants) | 40 | 19
  Week 4/5 | 270943 [252682 to 289203] | 264155 [235979 to 292332]
  Week 10/12: number analyzed (Participants) | 40 | 19
  Week 10/12 | 247323 [230033 to 264612] | 261184 [231331 to 291038]

19. Secondary Outcome: Change in Platelet Counts From Entry
Description: as for outcome 13
Time Frame: Entry, Weeks 1, 2, 4, 5, 10, and 12
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: Platelets/mm^3
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
Platelets/mm^3
  Change From Entry to Week 1/2: number analyzed (Participants) | 40 | 18
  Change From Entry to Week 1/2 | 43018 [30682 to 55353] | 5264 [-13341 to 23868]
  Change From Entry to Week 4/5: number analyzed (Participants) | 40 | 18
  Change From Entry to Week 4/5 | 32435 [19716 to 45154] | 4603 [-11880 to 21086]
  Change From Entry to Week 10/12: number analyzed (Participants) | 40 | 18
  Change From Entry to Week 10/12 | 8815 [301 to 17329] | 3439 [-13976 to 20853]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in platelet values from Entry to Week 1/2; Test type: Superiority; p < 0.001, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 37754, 90% CI 2-sided [19609 to 55898] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in platelet values from Entry to Week 4/5; Test type: Superiority; p = 0.012, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 27832, 90% CI 2-sided [9849 to 45815] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 3: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in platelet values from Entry to Week 10/12; Test type: Superiority; p = 0.52, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 5376, 90% CI 2-sided [-8592 to 19344] — No Study Treatment mean

20. Secondary Outcome: Aspartate Aminotransferase (AST) (SGOT)
Description: as for outcome 12
Time Frame: Entry, Weeks 1, 2, 4, 5, 10, and 12
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
U/L
  Entry | 23.2 [20.6 to 25.7] | 23.1 [19.2 to 26.9]
  Week 1/2: number analyzed (Participants) | 40 | 19
  Week 1/2 | 28.2 [24.1 to 32.2] | 23.5 [18.1 to 28.9]
  Week 4/5: number analyzed (Participants) | 40 | 19
  Week 4/5 | 29.1 [25.2 to 32.9] | 21.2 [18.5 to 23.9]
  Week 10/12: number analyzed (Participants) | 40 | 19
  Week 10/12 | 24.7 [22.0 to 27.3] | 21.0 [18.2 to 23.8]

21. Secondary Outcome: Change in Aspartate Aminotransferase (AST) (SGOT) Values From Entry
Description: as for outcome 13
Time Frame: Entry, Weeks 1, 2, 4, 5, 10, and 12
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
U/L
  Change From Entry to Week 1/2: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 1/2 | 5.01 [2.17 to 7.86] | 0.05 [-4.35 to 4.45]
  Change From Entry to Week 4/5: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 4/5 | 5.89 [3.16 to 8.61] | -2.26 [-5.32 to 0.79]
  Change From Entry to Week 10/12: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 10/12 | 1.48 [-0.45 to 3.40] | -2.47 [-5.58 to 0.63]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in Aspartate Aminotransferase (AST) (SGOT) values from Entry to Week 1/2; Test type: Superiority; p = 0.05, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 4.96, 90% CI 2-sided [0.78 to 9.14] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in Aspartate Aminotransferase (AST) (SGOT) values from Entry to Week 4/5; Test type: Superiority; p < 0.001, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 8.15, 90% CI 2-sided [4.47 to 11.8] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 3: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in Aspartate Aminotransferase (AST) (SGOT) values from Entry to Week 10/12; Test type: Superiority; p = 0.025, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 3.95, 90% CI 2-sided [1.08 to 6.81] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

22. Secondary Outcome: Alanine Aminotransferase (ALT) (SGPT)
Description: as for outcome 12
Time Frame: Entry, Weeks 1, 2, 4, 5, 10, and 12
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
U/L
  Entry | 24.3 [21.0 to 27.6] | 26.9 [20.2 to 33.5]
  Week 1/2: number analyzed (Participants) | 40 | 19
  Week 1/2 | 28.5 [24.5 to 32.6] | 26.5 [18.7 to 34.2]
  Week 4/5: number analyzed (Participants) | 40 | 19
  Week 4/5 | 30.6 [24.9 to 36.2] | 22.4 [18.1 to 26.7]
  Week 10/12: number analyzed (Participants) | 40 | 19
  Week 10/12 | 24.9 [21.7 to 28.2] | 23.2 [18.6 to 27.7]

23. Secondary Outcome: Change in Alanine Aminotransferase (ALT) (SGPT) Values From Entry
Description: as for outcome 13
Time Frame: Entry, Weeks 1, 2, 4, 5, 10, and 12
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
U/L
  Change From Entry to Week 1/2: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 1/2 | 4.21 [1.62 to 6.81] | -0.68 [-3.30 to 1.94]
  Change From Entry to Week 4/5: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 4/5 | 6.25 [1.61 to 10.9] | -4.74 [-9.45 to -0.03]
  Change From Entry to Week 10/12: number analyzed (Participants) | 40 | 19
  Change From Entry to Week 10/12 | 0.64 [-1.72 to 2.99] | -4.00 [-8.52 to 0.52]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in Alanine Aminotransferase (ALT) (SGPT) values from Entry to Week 1/2; Test type: Superiority; p = 0.020, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 4.90, 90% CI 2-sided [1.46 to 8.33] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in Alanine Aminotransferase (ALT) (SGPT) values from Entry to Week 4/5; Test type: Superiority; p = 0.004, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 11.0, 90% CI 2-sided [4.84 to 17.1] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 3: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in Alanine Aminotransferase (ALT) (SGPT) values from Entry to Week 10/12; Test type: Superiority; p = 0.043, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 4.64, 90% CI 2-sided [0.88 to 8.39] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

24. Secondary Outcome: Fold Change in the Level of Plasma Interleukin 6 (IL-6)
Description: All values were log10 transformed prior to calculating change and conducting analyses and back transformed for presentation.
  Baseline is defined as the geometric mean of the Pre-entry and Entry values. Week 4/5 is defined as the geometric mean of the Week 4 and Week 5 values. Week 10/12 is defined as the geometric mean of the Week 10 and Week 12 values. Fold change was calculated as the value at Week 10/12 divided by the value at Baseline and the value at Week 4/5 divided by the value at Week 10/12.
Time Frame: Pre-entry, Entry, Weeks 4, 5, 10 and 12
Population: As-treated population w/ results at each time point (data at baseline and week 4/5; for the Ruxolitinib arm, remained on study treatment through week 4/5 and missed no more than 6 doses cumulatively; did not change ART, use prohibited medications, or have confirmed virologic failure through week 4/5; not found to be ineligible after randomization).
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 36 | 17
Fold Change
  Fold Change from Baseline to Week 10/12 | 1.16 [0.96 to 1.41] | 1.06 [0.82 to 1.36]
  Fold Change from Week 4/5 to Week 10/12 | 1.26 [1.06 to 1.49] | 0.92 [0.76 to 1.11]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Plasma Interleukin 6 (IL-6) from baseline to Week 10/12; Test type: Superiority; p = 0.56, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.10, 90% CI 2-sided [0.84 to 1.44] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Plasma Interleukin 6 (IL-6) from Week 4/5 to Week 10/12; Test type: Superiority; p = 0.026, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.37, 90% CI 2-sided [1.09 to 1.73] — [estimate comment as in outcome 5, analysis 1]

25. Secondary Outcome: Fold Change in the Level of Soluble CD14 (sCD14)
Description: All values were log10 transformed prior to calculating change and conducting analyses and back transformed for presentation.
  Baseline is defined as the geometric mean of the Pre-entry and Entry values. Week 4/5 is defined as the geometric mean of the Week 4 and Week 5 values. Fold change was calculated as the value at Week 4/5 divided by the value at Baseline, the value at Week 12 divided by the value at Baseline, and the value at Week 12 divided by the value at Week 4/5.
Time Frame: Pre-entry, Entry, Weeks 4, 5, and 12
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 37 | 18
Fold Change
  Fold Change from Baseline to Week 4/5 | 0.96 [0.90 to 1.02] | 1.08 [0.93 to 1.26]
  Fold Change from Baseline to Week 12: number analyzed (Participants) | 35 | 17
  Fold Change from Baseline to Week 12 | 1.02 [0.91 to 1.15] | 1.08 [0.93 to 1.25]
  Fold Change from Week 4/5 to Week 12: number analyzed (Participants) | 35 | 17
  Fold Change from Week 4/5 to Week 12 | 1.08 [0.96 to 1.20] | 1.02 [0.86 to 1.21]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in soluble CD14 (sCD14) from baseline to Week 4/5; Test type: Superiority; p = 0.07, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.89, 90% CI 2-sided [0.80 to 0.99] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in soluble CD14 (sCD14) from baseline to Week 12; Test type: Superiority; p = 0.59, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.95, 90% CI 2-sided [0.80 to 1.12] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in soluble CD14 (sCD14) from Week 4/5 to Week 12; Test type: Superiority; p = 0.56, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.06, 90% CI 2-sided [0.90 to 1.24] — [estimate comment as in outcome 5, analysis 1]

26. Secondary Outcome: Change in CD4+ T Cell Count
Description: Baseline is defined as the average of pre-entry and entry. Absolute change was calculated as the value at Week 2 minus the value at Baseline, the value at week 5 minus the value at baseline, the value at week 12 minus the value at baseline, and the value at week 5 minus the value at week 12.
Time Frame: Pre-entry, Entry, Weeks 2, 5, and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 37 | 18
cells/mm^3
  Change from Baseline to Week 2 | 131.2 [66.6 to 195.8] | -10.9 [-75.0 to 53.3]
  Change from Baseline to Week 5: number analyzed (Participants) | 36 | 18
  Change from Baseline to Week 5 | 66.1 [0.87 to 131.2] | -8.19 [-64.1 to 47.7]
  Change from Baseline to Week 12: number analyzed (Participants) | 35 | 18
  Change from Baseline to Week 12 | 3.27 [-76.4 to 82.9] | 42.2 [-45.6 to 130.0]
  Change from Week 5 to Week 12: number analyzed (Participants) | 35 | 18
  Change from Week 5 to Week 12 | -62.1 [-153 to 28.9] | 50.4 [-46.2 to 146.9]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in CD4+ T cell counts from Baseline to Week 2; Test type: Superiority; p = 0.007, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 142.1, 90% CI 2-sided [57.6 to 227] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in CD4+ T cell counts from Baseline to Week 5; Test type: Superiority; p = 0.14, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 74.3, 90% CI 2-sided [-8.23 to 156.7] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 3: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in CD4+ T cell counts from Baseline to Week 12; Test type: Superiority; p = 0.54, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -38.9, 90% CI 2-sided [-143 to 65.5] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 4: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; There is no difference between the two arms in the change in CD4+ T cell counts from Week 5 to Week 12; Test type: Superiority; p = 0.12, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -112, 90% CI 2-sided [-231 to 5.90] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

27. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA Level Above the Limit of Quantification
Description: Participants were required to be virally suppressed, with a plasma HIV-1 RNA level below 40 copies/mL. The number of participants with plasma HIV-1 RNA level above the limit of quantification is reported at each time point.
Time Frame: Entry, Weeks 2, 5, and 12
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
Participants
  Entry | 1 | 0
  Week 2: number analyzed (Participants) | 40 | 19
  Week 2 | 0 | 0
  Week 5: number analyzed (Participants) | 40 | 19
  Week 5 | 2 | 0
  Week 12: number analyzed (Participants) | 40 | 19
  Week 12 | 1 | 0

28. Secondary Outcome: Relative Risks of HIV-1 RNA by Single Copy Assay (SCA) < 0.4 Copies/mL
Description: HIV-1 RNA was measured via Single Copy Assay Using Primer in Integrase (iSCA), results were reported as below or above the assay limit of detection (LOD) (LOD = 0.4 copies/mL). GEE models for binary data were used to calculate the relative risk of having HIV-1 RNA by iSCA <0.4 copies/mL (Week 5 compared to Entry, Week 12 compared to Entry, and Week 12 compared to Week 5).
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Relative Risk
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 37 | 18
Relative Risk
  Relative risk of SCA<LOD at Wk 5 compared to Entry: number analyzed (Participants) | 35 | 18
  Relative risk of SCA<LOD at Wk 5 compared to Entry | 1.20 [0.84 to 1.72] | 1.22 [0.82 to 1.81]
  Relative risk of SCA<LOD at Wk12 compared to Entry: number analyzed (Participants) | 35 | 18
  Relative risk of SCA<LOD at Wk12 compared to Entry | 0.82 [0.44 to 1.53] | 1.11 [0.64 to 1.92]
  Relative risk of SCA<LOD at Wk12 compared to Wk5: number analyzed (Participants) | 33 | 18
  Relative risk of SCA<LOD at Wk12 compared to Wk5 | 0.75 [0.43 to 1.32] | 0.91 [0.60 to 1.38]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in HIV-1 RNA by iSCA from Entry to Week 5; Test type: Superiority; p = 0.94, GEE — Not adjusted for multiple comparisons. Two-sided 10% alpha; A GEE model for binary data was used to compare changes in iSCA because a substantial proportion of data was below the assay limit; Risk Ratio (RR) = 0.98, 90% CI 2-sided [0.65 to 1.49] — Risk ratio is Ruxolitinib risk divided by No Study Treatment risk
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in HIV-1 RNA by iSCA from Entry to Week 12; Test type: Superiority; p = 0.46, GEE — Not adjusted for multiple comparisons. Two-sided 10% alpha; [statistical method as in outcome 28, analysis 1]; Risk Ratio (RR) = 0.74, 90% CI 2-sided [0.37 to 1.46] — Risk ratio is Ruxolitinib risk divided by No Study Treatment risk
Statistical Analysis 3: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in HIV-1 RNA by iSCA from Week 5 to Week 12; Test type: Superiority; p = 0.59, GEE — Not adjusted for multiple comparisons. Two-sided 10% alpha; [statistical method as in outcome 28, analysis 1]; Risk Ratio (RR) = 0.83, 90% CI 2-sided [0.46 to 1.48] — Risk ratio is Ruxolitinib risk divided by No Study Treatment risk

29. Secondary Outcome: Fold Change in the Level of Plasma Tumor Necrosis Factor Alpha (TNF Alpha)
Description: All values were log10 transformed prior to calculating change and conducting analyses and back transformed for presentation.
  Fold change was calculated as the value at Week 5 divided by the value at Entry and the value at Week 12 divided by the value at Entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 36 | 17
Fold Change
  Fold Change from Entry to Week 5 | 0.79 [0.71 to 0.88] | 0.90 [0.82 to 0.99]
  Fold Change from Entry to Week 12: number analyzed (Participants) | 34 | 17
  Fold Change from Entry to Week 12 | 0.85 [0.63 to 1.14] | 0.92 [0.73 to 1.15]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Tumor Necrosis Factor alpha (TNF alpha) from entry to Week 5; Test type: Superiority; p = 0.11, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.88, 90% CI 2-sided [0.76 to 1.01] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Tumor Necrosis Factor alpha (TNF alpha) from entry to Week 12; Test type: Superiority; p = 0.71, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.92, 90% CI 2-sided [0.64 to 1.33] — [estimate comment as in outcome 5, analysis 1]

30. Secondary Outcome: Fold Change in the Level of Plasma Interleukin 1 Beta (IL-1 Beta)
Description: as for outcome 29
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 36 | 17
Fold Change
  Fold Change from Entry to Week 5 | 0.96 [0.72 to 1.27] | 0.75 [0.55 to 1.03]
  Fold Change from Entry to Week 12: number analyzed (Participants) | 34 | 17
  Fold Change from Entry to Week 12 | 1.24 [0.60 to 2.60] | 0.78 [0.28 to 2.21]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Interleukin 1 beta (IL-1 beta) from entry to Week 5; Test type: Superiority; p = 0.30, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.27, 90% CI 2-sided [0.87 to 1.86] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Interleukin 1 beta (IL-1 beta) from entry to Week 12; Test type: Superiority; p = 0.46, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.59, 90% CI 2-sided [0.56 to 4.49] — [estimate comment as in outcome 5, analysis 1]

31. Secondary Outcome: Fold Change in the Level of Plasma Interleukin 7 (IL-7)
Description: as for outcome 29
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 36 | 17
Fold Change
  Fold Change from Entry to Week 5 | 1.04 [0.82 to 1.33] | 0.81 [0.55 to 1.18]
  Fold Change from Entry to Week 12: number analyzed (Participants) | 34 | 17
  Fold Change from Entry to Week 12 | 1.23 [0.92 to 1.65] | 1.04 [0.76 to 1.42]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Interleukin 7 (IL-7) from entry to Week 5; Test type: Superiority; p = 0.24, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.29, 90% CI 2-sided [0.90 to 1.84] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Interleukin 7 (IL-7) from entry to Week 12; Test type: Superiority; p = 0.46, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.19, 90% CI 2-sided [0.81 to 1.74] — [estimate comment as in outcome 5, analysis 1]

32. Secondary Outcome: Fold Change in the Level of Interleukin 1 Alpha (IL-1 Alpha)
Description: Laboratory testing was not performed so the data are not available.
Time Frame: Pre-entry, Entry, Weeks 4, 5, and 12
Population: Results not reported.
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Fold Change in the Level of Interferon Gamma-induced Protein 10 (IP-10)
Description: Laboratory testing was not performed so the data are not available.
Time Frame: Pre-entry, Entry, Weeks 4, 5, and 12
Population: Results not reported.
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Fold Change in the Level of Macrophage Colony-stimulating Factor
Description: Laboratory testing was not performed so the data are not available.
Time Frame: Pre-entry, Entry, Weeks 4, 5, and 12
Population: Results not reported.
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Fold Change in the Level of Neopterin
Description: Data not available because the testing lab reported that the values were unreliable.
Time Frame: Pre-entry, Entry, Weeks 4, 5, and 12
Population: Results not reported.
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Fold Change in the Level of Plasma Interleukin 10 (IL-10)
Description: as for outcome 29
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 35 | 17
Fold Change
  Fold Change from Entry to Week 5 | 0.94 [0.75 to 1.17] | 0.82 [0.47 to 1.43]
  Fold Change from Entry to Week 12: number analyzed (Participants) | 34 | 17
  Fold Change from Entry to Week 12 | 0.65 [0.37 to 1.15] | 0.67 [0.39 to 1.16]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Interleukin 10 (IL-10) from entry to Week 5; Test type: Superiority; p = 0.56, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.15, 90% CI 2-sided [0.77 to 1.72]; Mean difference is Ruxolitinib geometric mean minus No Study Treatment geometric mean. All values were log10 transformed prior to calculating change and conducting analyses and back transformed for presentation
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Interleukin 10 (IL-10) from entry to Week 12; Test type: Superiority; p = 0.95, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.97, 90% CI 2-sided [0.47 to 2.01] — [estimate comment as in outcome 5, analysis 1]

37. Secondary Outcome: Fold Change in the Level of Plasma Interleukin 15 (IL-15)
Description: as for outcome 29
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 36 | 17
Fold Change
  Fold Change from Entry to Week 5 | 1.33 [1.19 to 1.48] | 0.99 [0.87 to 1.13]
  Fold Change from Entry to Week 12: number analyzed (Participants) | 34 | 17
  Fold Change from Entry to Week 12 | 1.06 [0.88 to 1.27] | 0.98 [0.87 to 1.11]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in TInterleukin 15 (IL-15) from entry to Week 5; Test type: Superiority; p = 0.002, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.34, 90% CI 2-sided [1.15 to 1.56] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in TInterleukin 15 (IL-15) from entry to Week 12; Test type: Superiority; p = 0.60, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.07, 90% CI 2-sided [0.86 to 1.34] — [estimate comment as in outcome 5, analysis 1]

38. Secondary Outcome: Fold Change in the Level of Plasma Interleukin 18 (IL-18)
Description: as for outcome 29
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 36 | 17
Fold Change
  Fold Change from Entry to Week 5 | 0.89 [0.81 to 0.98] | 0.95 [0.84 to 1.07]
  Fold Change from Entry to Week 12: number analyzed (Participants) | 34 | 17
  Fold Change from Entry to Week 12 | 1.05 [0.88 to 1.24] | 1.02 [0.90 to 1.15]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Interleukin 18 (IL-18) from entry to Week 5; Test type: Superiority; p = 0.40, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.94, 90% CI 2-sided [0.82 to 1.07] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Interleukin 18 (IL-18) from entry to Week 12; Test type: Superiority; p = 0.82, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.03, 90% CI 2-sided [0.83 to 1.27] — [estimate comment as in outcome 5, analysis 1]

39. Secondary Outcome: Fold Change in the Level of Plasma Transforming Growth Factor Beta 1 (TGF Beta-1)
Description: as for outcome 29
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 36 | 17
Fold Change
  Fold Change from Entry to Week 5 | 0.90 [0.74 to 1.11] | 0.60 [0.44 to 0.83]
  Fold Change from Entry to Week 12: number analyzed (Participants) | 34 | 17
  Fold Change from Entry to Week 12 | 1.91 [0.86 to 4.22] | 0.93 [0.71 to 1.24]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Transforming Growth Factor beta 1 (TGF beta-1) from entry to Week 5; Test type: Superiority; p = 0.028, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.50, 90% CI 2-sided [1.11 to 2.02] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Transforming Growth Factor beta 1 (TGF beta-1) from entry to Week 12; Test type: Superiority; p = 0.21, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 2.04, 90% CI 2-sided [0.79 to 5.25] — [estimate comment as in outcome 5, analysis 1]

40. Secondary Outcome: Fold Change in the Level of Plasma Transforming Growth Factor Beta 2 (TGF Beta-2)
Description: as for outcome 29
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 36 | 17
Fold Change
  Fold Change from Entry to Week 5 | 0.96 [0.81 to 1.13] | 0.69 [0.52 to 0.90]
  Fold Change from Entry to Week 12: number analyzed (Participants) | 34 | 17
  Fold Change from Entry to Week 12 | 0.90 [0.49 to 1.65] | 0.94 [0.62 to 1.41]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Transforming Growth Factor beta 2 (TGF beta-2) from entry to Week 5; Test type: Superiority; p = 0.031, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.39, 90% CI 2-sided [1.08 to 1.79] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Transforming Growth Factor beta 2 (TGF beta-2) from entry to Week 12; Test type: Superiority; p = 0.93, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.96, 90% CI 2-sided [0.46 to 2.02] — [estimate comment as in outcome 5, analysis 1]

41. Secondary Outcome: Fold Change in the Level of Plasma Transforming Growth Factor Beta 3 (TGF Beta-3)
Description: as for outcome 29
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 36 | 17
Fold Change
  Fold Change from Entry to Week 5 | 0.99 [0.52 to 1.90] | 0.63 [0.23 to 1.69]
  Fold Change from Entry to Week 12: number analyzed (Participants) | 33 | 17
  Fold Change from Entry to Week 12 | 0.67 [0.39 to 1.16] | 0.99 [0.42 to 2.36]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Transforming Growth Factor beta 3 (TGF beta-3) from entry to Week 5; Test type: Superiority; p = 0.43, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.57, 90% CI 2-sided [0.61 to 4.05] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Transforming Growth Factor beta 3 (TGF beta-3) from entry to Week 12; Test type: Superiority; p = 0.41, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.68, 90% CI 2-sided [0.30 to 1.50] — [estimate comment as in outcome 5, analysis 1]

42. Secondary Outcome: Change in (CD3+CD4+) CD38+HLADR+
Description: Absolute change in the percent of parent cells (CD4+) that express CD38+HLADR+ cells (cellular marker of immune activation and inflammation in the peripheral blood).
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 34 | 17
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -0.27 [-0.47 to -0.07] | 0.08 [-0.18 to 0.33]
  Change from Entry to Week 12: number analyzed (Participants) | 33 | 16
  Change from Entry to Week 12 | 0.17 [0.01 to 0.32] | -0.10 [-0.38 to 0.18]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of CD38+HLADR+ among CD4+ T-cells from Entry to Week 5; Test type: Superiority; p = 0.038, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.34, 90% CI 2-sided [-0.61 to -0.07] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of CD38+HLADR+ among CD4+ T-cells from Entry to Week 12; Test type: Superiority; p = 0.07, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.27, 90% CI 2-sided [0.03 to 0.51] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

43. Secondary Outcome: Change in (CD3+CD8+) CD38+HLADR+
Description: Absolute change in the percent of parent cells (CD8+) that express CD38+HLADR+ cells (cellular marker of immune activation and inflammation in the peripheral blood).
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 34 | 17
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -1.16 [-1.67 to -0.65] | -0.28 [-1.09 to 0.53]
  Change from Entry to Week 12: number analyzed (Participants) | 33 | 16
  Change from Entry to Week 12 | 0.89 [0.16 to 1.62] | 0.03 [-0.94 to 1.00]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of CD38+HLADR+ among CD8+ T-cells from Entry to Week 5; Test type: Superiority; p = 0.05, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.88, 90% CI 2-sided [-1.62 to -0.13] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of CD38+HLADR+ among CD8+ T-cells from Entry to Week 12; Test type: Superiority; p = 0.16, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.86, 90% CI 2-sided [-0.16 to 1.88] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

44. Secondary Outcome: Change in (CD3+CD4+) CD25hi+
Description: Absolute change in the percent of parent cells (CD4+) that express CD25hi+ cells (cellular marker of immune activation and inflammation in the peripheral blood).
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 34 | 17
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -1.50 [-1.95 to -1.05] | 0.22 [-0.74 to 1.18]
  Change from Entry to Week 12: number analyzed (Participants) | 33 | 16
  Change from Entry to Week 12 | 0.08 [-0.37 to 0.53] | -0.08 [-0.79 to 0.62]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of CD25hi+ among CD4+ T-cells from Entry to Week 5; Test type: Superiority; p < 0.001, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -1.71, 90% CI 2-sided [-2.46 to -0.97] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of CD25hi+ among CD4+ T-cells from Entry to Week 12; Test type: Superiority; p = 0.68, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.16, 90% CI 2-sided [-0.50 to 0.82] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

45. Secondary Outcome: Change in (CD3+CD8+) CD25+
Description: Absolute change in the percent of parent cells (CD8+) that express CD25+ cells (cellular marker of immune activation and inflammation in the peripheral blood).
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 34 | 17
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -0.31 [-0.85 to 0.22] | -0.31 [-0.83 to 0.22]
  Change from Entry to Week 12: number analyzed (Participants) | 33 | 16
  Change from Entry to Week 12 | -0.53 [-1.25 to 0.19] | -0.38 [-1.23 to 0.48]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of CD25+ among CD8+ T-cells from Entry to Week 5; Test type: Superiority; p = 0.98, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.01, 90% CI 2-sided [-0.70 to 0.69] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of CD25+ among CD8+ T-cells from Entry to Week 12; Test type: Superiority; p = 0.79, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.16, 90% CI 2-sided [-1.13 to 0.82] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

46. Secondary Outcome: Change in (CD3+CD4+) CD127+
Description: Absolute change in the percent of parent cells (CD4+) that express CD127+ cells (cellular marker of immune activation and inflammation in the peripheral blood).
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 34 | 17
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | 2.65 [1.33 to 3.97] | -0.84 [-2.24 to 0.57]
  Change from Entry to Week 12: number analyzed (Participants) | 33 | 16
  Change from Entry to Week 12 | -1.48 [-2.94 to -0.03] | -0.19 [-1.97 to 1.60]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of CD127+ among CD4+ T-cells from Entry to Week 5; Test type: Superiority; p = 0.001, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 3.49, 90% CI 2-sided [1.75 to 5.22] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of CD127+ among CD4+ T-cells from Entry to Week 12; Test type: Superiority; p = 0.28, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -1.30, 90% CI 2-sided [-3.28 to 0.68]; Mean difference is Ruxolitinib mean minus No Study Treatment mean

47. Secondary Outcome: Change in (CD3+CD8+) CD127+
Description: Absolute change in the percent of parent cells (CD8+) that express CD127+ cells (cellular marker of immune activation and inflammation in the peripheral blood).
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 34 | 17
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | 5.42 [3.44 to 7.40] | -1.12 [-3.86 to 1.63]
  Change from Entry to Week 12: number analyzed (Participants) | 33 | 16
  Change from Entry to Week 12 | -0.09 [-2.53 to 2.35] | 0.11 [-3.05 to 3.26]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of CD127+ among CD8+ T-cells from Entry to Week 5; Test type: Superiority; p < 0.001, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 6.54, 90% CI 2-sided [3.76 to 9.31] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of CD127+ among CD8+ T-cells from Entry to Week 12; Test type: Superiority; p = 0.92, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.19, 90% CI 2-sided [-3.56 to 3.18] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

48. Secondary Outcome: Change in (CD3+CD4+) Ki67+
Description: Absolute change in the percent of parent cells (CD4+) that express Ki67+ cells (cellular marker of immune activation and inflammation in the peripheral blood).
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 34 | 17
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -0.26 [-0.55 to 0.02] | -0.19 [-0.95 to 0.58]
  Change from Entry to Week 12: number analyzed (Participants) | 33 | 16
  Change from Entry to Week 12 | 0.37 [0.00 to 0.73] | -0.39 [-1.11 to 0.32]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of Ki67+ among CD4+ T-cells from Entry to Week 5; Test type: Superiority; p = 0.82, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.07, 90% CI 2-sided [-0.61 to 0.47] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of Ki67+ among CD4+ T-cells from Entry to Week 12; Test type: Superiority; p = 0.033, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.76, 90% CI 2-sided [0.18 to 1.34] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

49. Secondary Outcome: Change in (CD3+CD8+) Ki67+
Description: Absolute change in the percent of parent cells (CD8+) that express Ki67+ cells (cellular marker of immune activation and inflammation in the peripheral blood).
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 34 | 17
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -0.64 [-0.88 to -0.41] | -0.65 [-1.50 to 0.19]
  Change from Entry to Week 12: number analyzed (Participants) | 33 | 16
  Change from Entry to Week 12 | 0.59 [-0.03 to 1.21] | 0.04 [-1.26 to 1.33]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of Ki67+ among CD8+ T-cells from Entry to Week 5; Test type: Superiority; p = 0.98, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.01, 90% CI 2-sided [-0.53 to 0.55] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of Ki67+ among CD8+ T-cells from Entry to Week 12; Test type: Superiority; p = 0.37, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.55, 90% CI 2-sided [-0.46 to 1.57] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

50. Secondary Outcome: Change in (CD3+CD4+) Bcl2+
Description: Absolute change in the percent of parent cells (CD4+) that express Bcl2+ cells (cellular marker of immune activation and inflammation in the peripheral blood).
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 34 | 17
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -3.77 [-4.93 to -2.62] | -0.48 [-1.31 to 0.35]
  Change from Entry to Week 12: number analyzed (Participants) | 33 | 16
  Change from Entry to Week 12 | -0.67 [-1.11 to -0.23] | 0.06 [-0.81 to 0.92]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of Bcl2+ among CD4+ T-cells from Entry to Week 5; Test type: Superiority; p < 0.001, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -3.30, 90% CI 2-sided [-4.72 to -1.87] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of Bcl2+ among CD4+ T-cells from Entry to Week 12; Test type: Superiority; p = 0.09, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.73, 90% CI 2-sided [-1.42 to -0.03] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

51. Secondary Outcome: Change in (CD3+CD8+) Bcl2+
Description: Absolute change in the percent of parent cells (CD8+) that express Bcl2+ cells (cellular marker of immune activation and inflammation in the peripheral blood).
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 34 | 17
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -5.64 [-7.19 to -4.09] | -0.24 [-1.20 to 0.72]
  Change from Entry to Week 12: number analyzed (Participants) | 33 | 16
  Change from Entry to Week 12 | -1.29 [-2.14 to -0.44] | -0.06 [-1.50 to 1.38]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of Bcl2+ among CD8+ T-cells from Entry to Week 5; Test type: Superiority; p < 0.001, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -5.40, 90% CI 2-sided [-7.29 to -3.50] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of Bcl2+ among CD8+ T-cells from Entry to Week 12; Test type: Superiority; p = 0.11, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -1.23, 90% CI 2-sided [-2.51 to 0.05] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

52. Secondary Outcome: Change in (CD3+CD4+) a4b7+
Description: Absolute change in the percent of parent cells (CD4+) that express a4b7+ cells (cellular marker of immune activation and inflammation in the peripheral blood).
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 34 | 17
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -2.16 [-3.43 to -0.88] | -0.62 [-3.64 to 2.40]
  Change from Entry to Week 12: number analyzed (Participants) | 33 | 16
  Change from Entry to Week 12 | -0.01 [-1.45 to 1.43] | 0.38 [-1.58 to 2.34]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of a4b7+ among CD4+ T-cells from Entry to Week 5; Test type: Superiority; p = 0.26, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -1.54, 90% CI 2-sided [-3.78 to 0.70] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of a4b7+ among CD4+ T-cells from Entry to Week 12; Test type: Superiority; p = 0.74, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.39, 90% CI 2-sided [-2.41 to 1.62] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

53. Secondary Outcome: Change in (CD3+CD8+) a4b7+
Description: Absolute change in the percent of parent cells (CD8+) that express a4b7+ cells (cellular marker of immune activation and inflammation in the peripheral blood).
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 34 | 17
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | 0.01 [-1.62 to 1.65] | -0.54 [-3.30 to 2.22]
  Change from Entry to Week 12: number analyzed (Participants) | 33 | 16
  Change from Entry to Week 12 | 0.91 [-0.80 to 2.61] | 0.59 [-1.99 to 3.18]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of a4b7+ among CD8+ T-cells from Entry to Week 5; Test type: Superiority; p = 0.71, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.55, 90% CI 2-sided [-1.90 to 3.00] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of a4b7+ among CD8+ T-cells from Entry to Week 12; Test type: Superiority; p = 0.83, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.31, 90% CI 2-sided [-2.15 to 2.78] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

54. Secondary Outcome: Change in (CD3+CD4+) CX3CR1+
Description: Absolute change in the percent of parent cells (CD4+) that express CX3CR1+ cells (cellular marker of immune activation and inflammation in the peripheral blood).
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 35 | 16
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -1.55 [-2.14 to -0.96] | -0.22 [-1.00 to 0.56]
  Change from Entry to Week 12 | -0.21 [-0.66 to 0.24] | -0.04 [-1.26 to 1.19]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of CX3CR1+ among CD4+ T-cells from Entry to Week 5; Test type: Superiority; p = 0.010, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -1.33, 90% CI 2-sided [-2.16 to -0.50] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in the expression of CX3CR1+ among CD4+ T-cells from Entry to Week 12; Test type: Superiority; p = 0.74, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.17, 90% CI 2-sided [-1.02 to 0.68] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

55. Secondary Outcome: Change in (CD3+CD8+) CX3CR1+
Description: Absolute change in the percent of parent cells (CD8+) that express CX3CR1+ cells (cellular marker of immune activation and inflammation in the peripheral blood).
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 35 | 16
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -4.31 [-5.46 to -3.16] | -1.07 [-3.71 to 1.57]
  Change from Entry to Week 12 | -0.39 [-1.79 to 1.02] | -0.22 [-2.87 to 2.43]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; [analysis description as in outcome 43, analysis 1]; Test type: Superiority; p = 0.008, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -3.24, 90% CI 2-sided [-5.22 to -1.27] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; [analysis description as in outcome 43, analysis 2]; Test type: Superiority; p = 0.90, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Median Difference (Net) = -0.17, 90% CI 2-sided [-2.38 to 2.05] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

56. Secondary Outcome: Change in CD69
Description: Data not available because the team decided they were no longer clinically relevant, so samples were not tested for CD69.
Time Frame: Entry, Weeks 5 and 12
Population: Results not reported.
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 0 | 0

57. Secondary Outcome: Change in PAR-1
Description: Data not available because the team decided they were no longer clinically relevant, so samples were not tested for PAR-1.
Time Frame: Entry, Weeks 5 and 12
Population: Results not reported.
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 0 | 0

58. Secondary Outcome: Change in Classical Monocytes (CD14+CD16-)
Description: Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 35 | 16
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | 0.95 [-1.49 to 3.40] | -0.43 [-2.66 to 1.80]
  Change from Entry to Week 12 | 1.15 [-0.85 to 3.15] | -1.06 [-4.27 to 2.15]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in classical monocytes (CD14+CD16-) from Entry to Week 5; Test type: Superiority; p = 0.47, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.39, 90% CI 2-sided [-1.83 to 4.61] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in classical monocytes (CD14+CD16-) from Entry to Week 12; Test type: Superiority; p = 0.22, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 2.21, 90% CI 2-sided [-0.77 to 5.18] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

59. Secondary Outcome: Change in Classical Monocytes (CD14+CD16-) Expressing CD163+
Description: Absolute change in the percent of classical monocytes (CD14+CD16-) that express CD163+.
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 35 | 16
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -1.16 [-5.47 to 3.15] | 3.18 [-4.62 to 11.0]
  Change from Entry to Week 12 | -5.05 [-9.68 to -0.43] | 4.76 [-2.36 to 11.9]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in classical monocytes (CD14+CD16-) expressing CD163+ from Entry to Week 5; Test type: Superiority; p = 0.28, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -4.34, 90% CI 2-sided [-11.0 to 2.35] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in classical monocytes (CD14+CD16-) expressing CD163+ from Entry to Week 12; Test type: Superiority; p = 0.019, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -9.81, 90% CI 2-sided [-16.6 to -3.02] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

60. Secondary Outcome: Change in Classical Monocytes (CD14+CD16-) Expressing CCR2+
Description: Absolute change in the percent of classical monocytes (CD14+CD16-) that express CCR2+.
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 35 | 16
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -1.24 [-2.83 to 0.35] | -0.43 [-2.44 to 1.58]
  Change from Entry to Week 12 | -0.84 [-1.77 to 0.09] | 0.86 [-1.43 to 3.15]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in classical monocytes (CD14+CD16-) expressing CCR2+ from Entry to Week 5; Test type: Superiority; p = 0.55, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.81, 90% CI 2-sided [-3.02 to 1.41] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in classical monocytes (CD14+CD16-) expressing CCR2+ from Entry to Week 12; Test type: Superiority; p = 0.09, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -1.70, 90% CI 2-sided [-3.36 to -0.04] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

61. Secondary Outcome: Change in Classical Monocytes (CD14+CD16-) Expressing CX3CR1+
Description: Absolute change in the percent of classical monocytes (CD14+CD16-) that express CX3CR1+.
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 35 | 16
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -1.72 [-2.99 to -0.44] | -0.25 [-1.52 to 1.02]
  Change from Entry to Week 12 | -0.62 [-2.89 to 1.65] | 1.00 [-0.96 to 2.96]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in classical monocytes (CD14+CD16-) expressing CX3CR1+ from Entry to Week 5; Test type: Superiority; p = 0.15, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -1.47, 90% CI 2-sided [-3.17 to 0.23] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in classical monocytes (CD14+CD16-) expressing CX3CR1+ from Entry to Week 12; Test type: Superiority; p = 0.37, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -1.62, 90% CI 2-sided [-4.59 to 1.35] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

62. Secondary Outcome: Change in Inflammatory Monocytes (CD14+CD16+)
Description: as for outcome 58
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 35 | 16
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -1.21 [-2.46 to 0.03] | -0.36 [-1.57 to 0.86]
  Change from Entry to Week 12 | -0.49 [-1.85 to 0.88] | 0.22 [-1.44 to 1.88]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in inflammatory monocytes (CD14+CD16+) from Entry to Week 5; Test type: Superiority; p = 0.39, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.86, 90% CI 2-sided [-2.51 to 0.80] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in inflammatory monocytes (CD14+CD16+) from Entry to Week 12; Test type: Superiority; p = 0.54, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.70, 90% CI 2-sided [-2.59 to 1.19] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

63. Secondary Outcome: Change in Inflammatory Monocytes (CD14+CD16+) Expressing CD163+
Description: Absolute change in the percent of inflammatory monocytes (CD14+CD16-) that express CD163+.
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 35 | 16
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -3.88 [-8.29 to 0.53] | 2.14 [-2.62 to 6.89]
  Change from Entry to Week 12 | -4.40 [-7.97 to -0.82] | 2.00 [-1.00 to 4.99]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in inflammatory monocytes (CD14+CD16+) expressing CD163+ from Entry to Week 5; Test type: Superiority; p = 0.10, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -6.02, 90% CI 2-sided [-12.0 to -0.06] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in inflammatory monocytes (CD14+CD16+) expressing CD163+ from Entry to Week 12; Test type: Superiority; p = 0.026, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -6.39, 90% CI 2-sided [-11.1 to -1.73] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

64. Secondary Outcome: Change in Inflammatory Monocytes (CD14+CD16+) Expressing CCR2+
Description: Absolute change in the percent of inflammatory monocytes (CD14+CD16+) that express CCR2+.
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 35 | 16
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | 2.95 [-1.81 to 7.71] | 2.67 [-6.40 to 11.7]
  Change from Entry to Week 12 | -1.99 [-7.17 to 3.20] | 2.11 [-8.76 to 13.0]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in inflammatory monocytes (CD14+CD16+) expressing CCR2+ from Entry to Week 5; Test type: Superiority; p = 0.95, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.28, 90% CI 2-sided [-7.26 to 7.82] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in inflammatory monocytes (CD14+CD16+) expressing CCR2+ from Entry to Week 12; Test type: Superiority; p = 0.43, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -4.10, 90% CI 2-sided [-12.6 to 4.45] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

65. Secondary Outcome: Change in Inflammatory Monocytes (CD14+CD16+) Expressing CX3CR1+
Description: Absolute change in the percent of inflammatory monocytes (CD14+CD16+) that express CX3CR1+.
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 35 | 16
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -4.38 [-8.56 to -0.20] | -5.61 [-12.6 to 1.40]
  Change from Entry to Week 12 | 0.58 [-5.47 to 6.63] | -3.18 [-7.12 to 0.76]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in inflammatory monocytes (CD14+CD16+) expressing CX3CR1+ from Entry to Week 5; Test type: Superiority; p = 0.74, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.23, 90% CI 2-sided [-5.08 to 7.54] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in inflammatory monocytes (CD14+CD16+) expressing CX3CR1+ from Entry to Week 12; Test type: Superiority; p = 0.42, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 3.76, 90% CI 2-sided [-3.94 to 11.5] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

66. Secondary Outcome: Change in Patrolling Monocytes (CD14dimCD16+)
Description: as for outcome 58
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 35 | 16
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | 0.20 [-1.56 to 1.96] | 0.83 [-0.98 to 2.65]
  Change from Entry to Week 12 | -0.70 [-2.28 to 0.89] | 0.87 [-1.69 to 3.42]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in patrolling monocytes (CD14dimCD16+) from Entry to Week 5; Test type: Superiority; p = 0.66, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -0.63, 90% CI 2-sided [-2.99 to 1.73] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in patrolling monocytes (CD14dimCD16+) from Entry to Week 12; Test type: Superiority; p = 0.27, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -1.56, 90% CI 2-sided [-3.93 to 0.80] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

67. Secondary Outcome: Change in Patrolling Monocytes (CD14dimCD16+) Expressing CD163+
Description: Absolute change in the percent of patrolling monocytes (CD14dimCD16+) that express CD163+.
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 35 | 16
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -4.05 [-7.55 to -0.54] | 3.05 [-0.27 to 6.37]
  Change from Entry to Week 12 | -1.09 [-5.90 to 3.73] | 0.41 [-5.06 to 5.88]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in patrolling monocytes (CD14dimCD16+) expressing CD163+ from Entry to Week 5; Test type: Superiority; p = 0.013, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -7.10, 90% CI 2-sided [-11.7 to -2.46] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in patrolling monocytes (CD14dimCD16+) expressing CD163+ from Entry to Week 12; Test type: Superiority; p = 0.70, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -1.49, 90% CI 2-sided [-8.06 to 5.07] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

68. Secondary Outcome: Change in Patrolling Monocytes (CD14dimCD16+) Expressing CCR2+
Description: Absolute change in the percent of patrolling monocytes (CD14dimCD16+) that express CCR2+.
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 35 | 16
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | 0.02 [-0.03 to 0.07] | 0.01 [-0.03 to 0.06]
  Change from Entry to Week 12 | 0.04 [-0.01 to 0.10] | 0.04 [-0.03 to 0.10]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in patrolling monocytes (CD14dimCD16+) expressing CCR2+ from Entry to Week 5; Test type: Superiority; p = 0.79, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.01, 90% CI 2-sided [-0.05 to 0.07] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in patrolling monocytes (CD14dimCD16+) expressing CCR2+ from Entry to Week 12; Test type: Superiority; p = 0.91, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.01, 90% CI 2-sided [-0.07 to 0.08] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

69. Secondary Outcome: Change in Patrolling Monocytes (CD14dimCD16+) Expressing CX3CR1+
Description: Absolute change in the percent of patrolling monocytes (CD14dimCD16+) that express CX3CR1+.
  Absolute change was calculated as the value at week 5 minus the value at entry, and the value at week 12 minus the value at entry.
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 24
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 35 | 16
Percent of Expression in Parent Cell
  Change from Entry to Week 5 | -5.48 [-9.38 to -1.59] | -2.64 [-9.44 to 4.17]
  Change from Entry to Week 12 | -2.39 [-7.64 to 2.87] | -2.42 [-4.73 to -0.10]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in patrolling monocytes (CD14dimCD16+) expressing CX3CR1+ from Entry to Week 5; Test type: Superiority; p = 0.43, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = -2.85, 90% CI 2-sided [-8.82 to 3.12] — Mean difference is Ruxolitinib mean minus No Study Treatment mean
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in patrolling monocytes (CD14dimCD16+) expressing CX3CR1+ from Entry to Week 12; Test type: Superiority; p = 0.99, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.03, 90% CI 2-sided [-6.53 to 6.60] — Mean difference is Ruxolitinib mean minus No Study Treatment mean

70. Secondary Outcome: Fold Change in Cellular HIV-1 DNA
Description: as for outcome 29
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 36 | 18
Fold Change
  Fold Change from Entry to Week 5 | 1.16 [0.96 to 1.41] | 0.62 [0.36 to 1.06]
  Fold Change from Entry to Week 12: number analyzed (Participants) | 34 | 17
  Fold Change from Entry to Week 12 | 1.18 [0.98 to 1.42] | 0.90 [0.52 to 1.55]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Cellular HIV-1 DNA from entry to Week 5; Test type: Superiority; p = 0.007, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Median Difference (Net) = 1.88, 90% CI 2-sided [1.29 to 2.73] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Cellular HIV-1 DNA from entry to Week 12; Test type: Superiority; p = 0.23, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.31, 90% CI 2-sided [0.90 to 1.90] — [estimate comment as in outcome 5, analysis 1]

71. Secondary Outcome: Fold Change in Cellular HIV-1 Total RNA
Description: as for outcome 29
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 36 | 18
Fold Change
  Fold Change from Entry to Week 5 | 1.06 [0.82 to 1.38] | 0.87 [0.66 to 1.15]
  Fold Change from Entry to Week 12: number analyzed (Participants) | 34 | 18
  Fold Change from Entry to Week 12 | 0.97 [0.74 to 1.29] | 0.95 [0.60 to 1.50]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in cellular HIV-1 total RNA from entry to Week 5; Test type: Superiority; p = 0.32, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.22, 90% CI 2-sided [0.87 to 1.72] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in cellular HIV-1 total RNA from entry to Week 12; Test type: Superiority; p = 0.91, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 1.03, 90% CI 2-sided [0.68 to 1.56] — [estimate comment as in outcome 5, analysis 1]

72. Secondary Outcome: Percentage of Participants With Detectable CMV Shedding
Description: Level of CMV shedding was summarized by study week and arm as the percentage of those above and below the assay limit of detection.
  Detectable CMV shedding was defined as CMV level > 0 copies/ml of elution. The percentage of participants with detectable CMV at any on-treatment time point (ever shedding at weeks 1, 2, 4, or 5) and any post-treatment time point (ever shedding at weeks 10 or 12) was contrasted between study arms.
Time Frame: Pre-entry, Entry, and Weeks 1, 2, 4, 5, 10, and 12
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 40 | 20
percentage of participants
  Pre-entry | 13 | 5
  Entry | 13 | 10
  Week 1 | 13 | 11
  Week 2: number analyzed (Participants) | 39 | 19
  Week 2 | 8 | 16
  Week 4: number analyzed (Participants) | 40 | 18
  Week 4 | 8 | 6
  Week 5: number analyzed (Participants) | 38 | 19
  Week 5 | 5 | 16
  Week 10: number analyzed (Participants) | 39 | 19
  Week 10 | 5 | 11
  Week 12: number analyzed (Participants) | 40 | 19
  Week 12 | 20 | 16
  Any Detectable CMV On-treatment: number analyzed (Participants) | 40 | 19
  Any Detectable CMV On-treatment | 18 | 26
  Any Detectable CMV Post-treatment: number analyzed (Participants) | 40 | 19
  Any Detectable CMV Post-treatment | 20 | 16
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the percentage of participants with detectable CMV at any on-treatment time point (ever shedding at weeks 1, 2, 4, or 5); Test type: Superiority; p = 0.40, Fisher Exact — Not adjusted for multiple comparisons. Two-sided 10% alpha; Fisher's Exact Mid P-Value
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the percentage of participants with detectable CMV at any post-treatment time point (ever shedding at weeks 10 or 12); Test type: Superiority; p = 0.87, Fisher Exact — Not adjusted for multiple comparisons. Two-sided 10% alpha; Fisher's Exact Mid P-Value

73. Secondary Outcome: Ruxolitinib Systemic Clearance (CL/F) From 2-compartment Pharmacokinetic (PK)
Description: Ruxolitinib plasma concentrations were fitted to a population 2-compartment distribution model, assuming first-order input, distribution and elimination from the plasma compartment, using nonlinear mixed-effects modeling software. We estimated parameter geometric means and proportional variabilities between subjects (IIV when feasible) and the variability in drug absorption between occasions (IOV week 1 and week 4/5), and related distribution volumes to body weight.
Time Frame: Week 1 and, Week 4/5; blood samples were drawn pre-dose and at 1-1.5, 2.5-4, 4-6, and 6-8 hours post-dosing
Population: Analysis was done on participants on the Ruxolitinib arm with intensive pharmacokinetic (PK) results. One participant was not included due to missing samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Arm A: Ruxolitinib
Number analyzed (Participants) | 39
L/hr | 14.5 (34)

74. Other Pre Specified Outcome: Change in 2 Long-terminal Repeat Sequences [LTRs]
Description: Data not available because all values were below assay limit.
Time Frame: Entry, Week 5, and Week 12
Population: Results not reported.
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 0 | 0

75. Other Pre Specified Outcome: Level of HHV Shedding (EBV, HSV, HHV-6, HHV-7, and HHV-8)
Description: Data not available because no samples were collected to test for these measures as the team decided they were no longer clinically relevant.
Time Frame: Pre-entry, Entry, Weeks 1, 2, 4, 5, 10, and 12
Population: Results not reported.
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 0 | 0

76. Other Pre Specified Outcome: Fold Change in Integrated DNA
Description: as for outcome 29
Time Frame: Entry, Weeks 5 and 12
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A: Ruxolitinib | Arm B: No Study Treatment
Number analyzed (Participants) | 33 | 17
Fold Change
  Fold Change from Entry to Week 5: number analyzed (Participants) | 33 | 16
  Fold Change from Entry to Week 5 | 1.10 [0.44 to 2.71] | 2.06 [0.61 to 6.98]
  Fold Change from Entry to Week 12: number analyzed (Participants) | 31 | 17
  Fold Change from Entry to Week 12 | 1.11 [0.31 to 4.00] | 1.20 [0.43 to 3.36]
Statistical Analysis 1: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Integrated DNA from entry to Week 5; Test type: Superiority; p = 0.40, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.53, 90% CI 2-sided [0.15 to 1.88] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Ruxolitinib vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the fold change in Integrated DNA from entry to Week 12; Test type: Superiority; p = 0.93, t-test, 2 sided — Not adjusted for multiple comparisons. Two-sided 10% alpha; 2-sample t-test with equal variance; Mean Difference (Net) = 0.92, 90% CI 2-sided [0.20 to 4.34] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: Week 0 to Week 12
Description: Protocol-defined recorded adverse events include: all diagnoses regardless of grade, Grade 2 or higher sign/symptoms and all non-traumatic bruising; Grade 2 or higher laboratory values and calculated creatinine clearance, creatinine, AST (SGOT), ALT (SGPT), ANC, hemoglobin, and platelet count regardless of grade; and any signs/symptoms or laboratory values that led to a change in treatment or met ICH, EAE, or SAE guidelines. The Division of AIDS AE Grading Table, Version 2.0 was used.
Groups:
- Ruxolitinib: Participants received ruxolitinib twice a day for 5 weeks. Participants were required to remain on ART regimen (not provided by the study) for the duration of the study.
  Ruxolitinib: 10 mg orally twice daily for 5 weeks
- No Study Treatment: Participants did not receive any study treatment. Participants were required to remain on ART regimen (not provided by the study) for the duration of the study.
Arm/Group | Ruxolitinib | No Study Treatment
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/40 | 0/20
Other Adverse Events (participants affected / at risk) | 31/40 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=40) | No Study Treatment (N=20)
Vitreous detachment (Eye disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=40) | No Study Treatment (N=20)
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Acute sinusitis (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 5 | 2
Aspartate aminotransferase increased (Investigations) | 8 | 2
Blood cholesterol increased (Investigations) | 9 | 7
Blood creatinine increased (Investigations) | 5 | 2
Blood glucose decreased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 7 | 3
Blood phosphorus decreased (Investigations) | 2 | 0
Blood triglycerides increased (Investigations) | 13 | 6
Low density lipoprotein increased (Investigations) | 7 | 8
Neutrophil count decreased (Investigations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-05-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT02475655/Prot_001.pdf
  • Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT02475655/SAP_000.pdf